CLINICAL TRIAL: NCT05319925
Title: Financial Effects of a Tumor Disease
Brief Title: Financial Effects of a Tumor Disease - Development and Validation of a Patient Reported Outcome Measure in Germany
Acronym: FIAT
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Chair of Methods in Empirical Social Research, Institute of Sociology, Technische Universität Dresden (Unknown); Health Economics and Health Care Management, Bielefeld University (Unknown); Haematology and Oncology, University of Jena (Unknown)
Responsible Party: Principal Investigator, Eva Winkler, MD, Prof. Dr. Dr., University Hospital Heidelberg
Other Study IDs: S-177/2021; 70113978 (Other Grant/Funding Number: German Cancer Aid)
Record Dates: First submitted 2022-02-08; First posted 2022-04-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Financial Toxicity; Financial Effects; Patient-reported Outcome; Cancer
MeSH Terms: conditions — Neoplasms; Financial Stress | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study 1: Initial examination of the developed questionnaire in the first 100 participants to identify problematic questions and to optimise the instrument.
  To evaluate test-retest reliability, collected data of the first 100 patients will be used as baseline value and re-assessed in Study 2.
  Interventions: Other: Patient reported outcome measure
- Study 2: Second examination in 300 additional participants and re-assessment in participants from Study 1 (n=400) to validate modified questionnaire in its final form.
  To evaluate test-retest reliability, data of Study 1 is compared against Study 2 of the same participant sample (n=100).
  Interventions: Other: Patient reported outcome measure

INTERVENTIONS:
Other: Patient reported outcome measure — Newly developed patient-reported instrument to measure financial effects of a cancer diagnosis and therapy of cancer patients in Germany
  Other Names: FIAT questionnaire

SUMMARY:
This study aims to develop and to validate a standardised German-language instrument for measuring experienced financial effects of a cancer diagnosis and therapy in a cross-sectional bi-centre study. Obtained data will make the patient-related description of financial difficulties more comprehensible, communicable and addressable in the future, e.g. by offering targeted advisory aids or considering financial effects in health technology assessments.

DETAILED DESCRIPTION:
Methods and analysis:

Phase 1: Construct definition and item generation

Preliminary study:

The preliminary study aims to identify dimensions, topics and risk factors that are relevant for the assessment of financial effects through qualitative interviews with patients, focus group discussions with potential users of a new instrument (social services, HTA-institutions, payers) and a systematic literature review.

Preliminary questionnaire:

In order to derive a pre-final questionnaire, the aim of this part of the study is to define the construct of financial effects and to generate a list of appropriate indicators for measuring financial effects based on the results available from the literature. The pre-final questionnaire will be peer-reviewed by the interdisciplinary project team (oncology/medical ethics, health economics, methods of empirical social research).

Phase 2: Questionnaire Piloting and Validation

Cognitive pre-test:

A cognitive pre-test of the pre-final questionnaire is conducted to examine comprehension of questions and response option and identify any potential problems respondents would have to understand the questions and to respond to them. The results are used in order to further optimize the first draft of the questionnaire.

Quantitative evaluation and validation:

Quantitative evaluation and validation of the developed questionnaire will be performed based on two studies on the target population by determining the distribution parameters of the indicators and their measurement characteristics. In the first study, the pre-final questionnaire will be tested and after adjustment, the final version will be applied in study 2. Participants of the first study (n=100) will be surveyed again within the second study (n=400 participants), while data of the additional participants (n=300) in study 2 will be measured at a single time point.

For validation purposes, additional scales measuring similar and unrelated constructs, as well as criteria (external concepts affected by financial effects) will be included in the questionnaire. Validity will be assessed by subsequent examining of different relationships between the developed instrument and predefined third variables and criteria. Factorial validity will be examined by factor analyses. Furthermore reliability and test-fairness of the instrument will be assessed through further psychometric testing.

Phase 3: Further applicability of the questionnaire To formulate well-founded recommendations for the use of the instrument, a pilot screening program for social services is evaluated through qualitative interviews with representatives of social services and patients regarding practicability of the instrument. A synthesis of all project results will translate into overall recommendations within the clinical and regulatory context.

ELIGIBILITY:
Inclusion Criteria:

* Any type of historically or cytological confirmed solid cancer or haematological malignancy with an ECOG-Status <2 and at least two month of cancer related therapy
* Patients are treated at the day care unit or ambulances of the NCT Heidelberg or oncological ward B100 at Jena University Hospital

Exclusion Criteria:

* Patients younger than 18 years old
* Patients who refuse or withdraw from informed consent
* No sufficient level of German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with all types of cancer who have undergone at least two months of cancer related therapy with an ECOG Status < 2, who are treated at the day care unit and ambulances of the NCT Heidelberg or conservative day care unit and oncological ward B100, Jena University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Validation of FIAT questionnaire (pre-version): Distribution analysis | 4 months
  Distribution analyses (correspondence to the normal distribution; skew and excess with evidence for possible ceiling and floor effects)
Validation of FIAT questionnaire (pre-version): Factorial validity | 4 months
  Exploratory Factor Analysis (EFA) will be used to analyse the factorial structure of the instrument to investigate which theoretically defined properties of the construct can adequately covered and differentiated with help of single indicators (items and questions).
Validation of FIAT questionnaire (pre-version): Reliability | 4 months
  Preliminary assessment of reliability with Guttmans-Lambda
Validation of FIAT questionnaire (final version): Distribution analysis | 5 months
  Distribution analyses (correspondence to the normal distribution; skew and excess with evidence for possible ceiling and floor effects)
Validation of FIAT questionnaire (final version): Factorial validity | 5 months
  Exploratory Factor Analysis (EFA) and Confirmatory Factor Analysis (CFA) will be used.
Validation of FIAT questionnaire (pre-version and final version): Test-retest-reliability | 5 months
  Correlations between the measurements between the first and second survey will be obtained to evaluate test-retest-reliability.
Validation of FIAT questionnaire (final version): Test-fairness | 5 months
  Test fairness will be evaluated by means of Multi-Group Confirmatory Factor Analysis (MG-CFA).

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Winkler, Prof. Dr. Dr., Principal Investigator — National Center for Tumor Diseases, University Hospital Heidelberg
Locations (1):
- National Center for Tumor Diseases, University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Pauge S, Surmann B, Mehlis K, Zueger A, Richter L, Menold N, Greiner W, Winkler EC. Patient-Reported Financial Distress in Cancer: A Systematic Review of Risk Factors in Universal Healthcare Systems. Cancers (Basel). 2021 Oct 7;13(19):5015. doi: 10.3390/cancers13195015. PMID 34638499
- [Derived] Zuger A, Mathies V, Mehlis K, Pauge S, Richter L, Surmann B, Ernst T, Menold N, Greiner W, Winkler E. Self-reported determinants for subjective financial distress: a qualitative interview study with German cancer patients. BMJ Open. 2025 Jan 28;15(1):e081432. doi: 10.1136/bmjopen-2023-081432. PMID 39880449
- See also: project description — https://www.nct-heidelberg.de/forschung/nct-core-services/nct-epoc/research/fiat.html